CLINICAL TRIAL: NCT00509418
Title: Efficacy and Safety of Viusid, a Nutritional Supplement, in Patients With Nonalcoholic Steatohepatitis. A Randomized, Controlled and Open Label Study
Brief Title: Efficacy and Safety of Viusid in Patients With Nonalcoholic Steatohepatitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Catalysis SL (Industry)
Responsible Party: Eduardo Vilar Gómez, National Institute of Gastroenterology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VIUNASH-07
Record Dates: First submitted 2007-07-30; First posted 2007-07-31 (Estimated); Last update posted 2009-01-12 (Estimated); Status verified 2009-01

CONDITIONS: Nonalcoholic Steatohepatitis
Keywords: Nonalcoholic steatohepatitis; Nonalcoholic Fatty Liver; Nutritional supplement; Diet; Exercise
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Motor Activity | interventions — Viusid; Dietary Supplements

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Viusid, a nutritional supplement, in combination with controlled diet and exercise
  Interventions: Dietary Supplement: Viusid
- B (Active Comparator): Controlled diet and exercise
  Interventions: Other: Hypocaloric Diet with controlled exercise

INTERVENTIONS:
Dietary Supplement: Viusid — Viusid, a nutritional supplement. Three oral sachets Daily 24 weeks
  Other Names: Nutritional supplement
  Arms: A
Other: Hypocaloric Diet with controlled exercise — Modified ADA diet in combination with controlled exercise daily 24 weeks
  Other Names: lifestyle modification
  Arms: B

SUMMARY:
The purpose of the study is to evaluate whether Viusid, a nutritional supplement, in combination with diet and exercise improve the histological results (steatosis, necro-inflammatory activity and fibrosis) in comparison with diet and exercise, during 24 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of steatohepatitis (minimal histological criteria for steatohepatitis include steatosis involving at least 5% of hepatocytes, lobular inflammation, and/or fibrosis)
* Age between 18 and 70 years
* Ability to provide informed consent
* Absence of significant alcohol ingestion (weekly ethanol consumption of less than 40 g)

Exclusion Criteria:

* Presence of other form of liver diseases (viral or autoimmune hepatitis, drug-induced liver disease, metabolic and hereditary liver disease and α-1 antitrypsin deficiency)
* Pregnancy or lactation
* Decompensated cirrhosis
* Presence of secondary cause of NAFL such as medications that induce steatosis (corticosteroids, estrogens, methotrexate, amiodarone, tamoxifen and calcium channel blockers) and gastrointestinal bypass surgery
* Pharmacological treatment with some potential benefit on NAFL including ursodeoxycholic acid, vitamin E, betaine, pioglitazone, rosiglitazone, metformin, pentoxifylline or gemfibrozil
* Fasting glucose levels greater than 250 mg per deciliter (13.3 mmol per liter)
* Contraindication to liver biopsy
* Refusal to participate in the study
* Concomitant disease with reduced life expectancy
* Severe psychiatric conditions
* Drug dependence

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2007-02; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
The histological improvement (steatosis, necro-inflammatory activity and fibrosis) at 24 weeks (end of the treatment). | 24 weeks

SECONDARY OUTCOMES:
Alanine aminotransferase levels (end of the treatment), δ-glutamyltransferase levels (end of the treatment), Body weight, Body Mass Index, Waist circumference (end of the treatment) Insulin resistance (HOMA) (end of the treatment) | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Adelaida Rodríguez de Miranda, MD, Principal Investigator — National Institute of Gastroenterology
Locations (1):
- National Institute of Gastroenterology, Vedado, La Habana, Cuba

REFERENCES:
- [Background] Vilar Gomez E, Gra Oramas B, Soler E, Llanio Navarro R, Ruenes Domech C. Viusid, a nutritional supplement, in combination with interferon alpha-2b and ribavirin in patients with chronic hepatitis C. Liver Int. 2007 Mar;27(2):247-59. doi: 10.1111/j.1478-3231.2006.01411.x. PMID 17311621